CLINICAL TRIAL: NCT02347969
Title: Evaluation of the Effect of the Dietary Supplement X34 on Skin Radiance of Healthy Volunteers With Dull Complexion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutratech Conseils (Other)
Collaborators: Research and Studies Center on the Integument (CERT) (Unknown); University of Franche-Comté (Other); Centre Hospitalier Universitaire de Besancon (Other); Clinical Investigation Center (CIC) INSERM 1431 (Unknown); INSERM UMR1098 (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DE-87; NCT02352415 (obsolete NCT alias)
Record Dates: First submitted 2015-01-16; First posted 2015-01-28 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Volunteers
Keywords: antioxidant; skin radiance; skin elasticity; skin firmness; skin hydration
MeSH Terms: interventions — 1,4-bis(3-carboxy-4-hydroxyphenylethenyl)-benzene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- X34 (Experimental): Arm supplemented with X34
  Interventions: Dietary Supplement: X34

INTERVENTIONS:
Dietary Supplement: X34 — Dietary supplement named X34

SUMMARY:
The main objective of this trial is to evaluate the effect of the daily dose of X34 dietary supplement on skin radiance (clinical assessment) for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female volunteers:
* Age: 40-70 years
* Who have a dull complexion evaluated by clinical scoring
* Phototype II to IV (annex 5)
* Non-smoking or smoking less than 5 cigarettes per day
* Did not change her eating habits, within one month before the start of the study and agreeing not change during the study
* With no history of facial skin care (peeling, mask…) 15 days before the beginning of the study and agreeing not to perform during the study
* Volunteers accepting not changing their local treatment on face
* Who agree to avoid UV exposure (sun or tanning booth) during the study
* Who have a fixed address and are entitled to Social Security or a similar National Insurance scheme
* Who sign a written informed consent

Exclusion Criteria:

* Pregnant, nursing, or intending to become pregnant in the course of the study
* With a history of allergy or hypersensitivity to the products or one of their components
* Having use oral nutritional supplements and/or vitamin supplementation less than one month before and/or refusing not consuming nutritional supplement during the study
* Having used cosmetics and/or topical preparations containing ingredients claiming efficacy on skin radiance less than 15 days before and/or during the study
* With a dermatosis, systemic disease or treatment susceptible to interfere with the evolution of the parameters of the study or with taking the nutritional supplement
* Participation in another clinical trial evaluating skin radiance during the last month before the study
* Participation in another clinical trial or volunteers being in the exclusion phase of such a trial, thus being unable to participate in any other one
* Who have forfeited their freedom by judiciary decision or are deemed legally incompetent
* Having perceived more than 4500 € as indemnification fees for participation in clinical trials during the preceding 12 months (including participation in this clinical trial)
* Unable to comply with the protocol constraints
* Who cannot be contacted by phone rapidly

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Skin radiance: clinical scoring | At 0 week and 8 weeks

SECONDARY OUTCOMES:
Subject self-assessments | At 0 week and 8 weeks
  Subjects will evaluate the radiance of their complexion by self-assessment.